CLINICAL TRIAL: NCT03446534
Title: The Norwegian Antibiotics for Pneumonia in Children Study
Acronym: NAPiC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Ostfold Hospital Trust (Other); Helse Stavanger HF (Other Government); Haukeland University Hospital (Other); Alesund Hospital (Other); St. Olavs Hospital (Other); Nordlandssykehuset HF (Other); University Hospital of North Norway (Other); University Hospital, Akershus (Other); Norwegian Institute of Public Health (Other Government); Klinbeforsk (Other)
Responsible Party: Principal Investigator, Håvard Ove Skjerven, Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/1863
Record Dates: First submitted 2018-02-17; First posted 2018-02-26 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Pneumonia Childhood; Lower Respiratory Tract Infection
Keywords: pneumonia; pre-school children; antibiotics; amoxicillin
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: The study is a phase IV double-blind, placebo-controlled, multicenter, nationwide, randomized superiority trial of amoxicillin versus placebo in children aged 1-5 years of age with a lower respiratory infection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxicillin (Experimental): Amoxicillin 100mg/ml mixture (Imacillin), 0.25ml/kg every 8 hours for 7 days.
  Interventions: Drug: Amoxicillin
- Placebo (Placebo Comparator): Placebo mixture 0.25ml/kg every 8 hours for 7 days
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Amoxicillin — Imacillin mixture
  Other Names: Imacillin
  Arms: Amoxicillin
Drug: Placebos — Placebo manufactured to mimic amoxicillin mixture (Imacillin)
  Arms: Placebo

SUMMARY:
This study evaluates the effect of amoxicillin in the treatment of lower airway infections in preschool children. Half of the patients will receive amoxicillin, while the other half will receive placebo.

DETAILED DESCRIPTION:
The overall objective of the study is to determine if antibiotic therapy is beneficial in children with pneumonia who do not have a highly suspicious bacterial infection, such as in lobar pneumonia.

Secondary objective is to determine whether antibiotic use influence the microbial flora, including antibiotic resistance, in the airways in the short or medium long term.

The study is a phase IV double-blind, placebo-controlled, multicenter, nationwide, randomized superiority trial of amoxicillin versus placebo in children aged 1-5 years of age with a lower respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-59 months
2. Fever:

   a. Temperature ≥ 38.0 at inclusion or reported within the last 24 hours
3. Tachypnoe, age specific 12-17mnd ≥ 46 breaths per minute 18-23mnd ≥ 40 breaths per minute 24-35mnd ≥ 34 breaths per minute 36-47mnd ≥ 29 breaths per minute 48-59mnd ≥ 27 breaths per minute
4. ≥ 1 sign of lower airway inflammation

   1. Cough (at inclusion or reported within the last 6 hours)
   2. Chest retractions (jugular, intercoastally or subcoastally)
   3. Grunting respiration
   4. Nasal flaring
   5. Crepitations by pulmonary auscultation
   6. Hypoxia (SpO2 ≤ 90%)
5. Weight between 6.0 and 28.0 kg. • Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations

Exclusion Criteria:

1. Clinical suspicion of bacterial pneumonia based upon a temperature ≥39.0°C and at least one of the following:

   1. Bronchial breathing sounds
   2. Unilaterally decreased breath sounds or unilateral percussion dullness
   3. Pulmonary lobar consolidation and/or radiological high suspicion of empyema on chest x-ray if this is obtained prior to inclusion in the trial.
2. Evidence of any bacterial infection requiring systemic antibiotics, including, but not exclusively:

   1. Clinical septicaemia
   2. Urinary tract infection
   3. Meningitis
3. Systemic antibiotics received within the last 7 days
4. Pulmonary lobar consolidation and/or radiological high suspicion of empyema on chest x-ray if this is obtained prior to inclusion in the trial.
5. History of any serious underlying disease that can increase the risk of bacterial pulmonary infections, including but not limited to:

   1. Haematological or oncological
   2. Immunodeficiency
   3. Congenital heart disease
   4. Neuromuscular impairment
   5. Development disorder, including Downs syndrome
   6. Bronchopulmonary dysplasia, cystic fibrosis, primary ciliary dyskinesia, poorly controlled asthma or other severe chronic lung diseases
6. Signs of lower obstructive airways with both of the following present by auscultation:

   1. prolonged expiration and
   2. generalised expiratory wheeze
7. Stridor by auscultation.
8. History of known or suspected adverse reactions to amoxicillin, or any other betalactam
9. Participating in another trial that might affect the current study
10. Any reason why, in the opinion of the investigator, the patient should not participate (e.g. not able to comply with study procedures)

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 884 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Therapy Failure | Within 7 days after inclusion
  Therapy failure as defined by attending physician, leading to end of intervention and administration of open-label antibiotics

SECONDARY OUTCOMES:
Thereapy failure leading to intravenous antibiotic therapy | Within 7 days after inclusion
  Therapy failure as defined by attending physician, leading to intravenous antibiotic therapy
Duration of fever | Up to 21 days after inclusion
  Duration of fever
Duration of symptoms of pneumonia | Up to 21 days after inclusion
  Duration of cough or respiratory distress (tachypnoe, retractions, grunting respiration or nasal flaring.

CONTACTS AND LOCATIONS:
Overall Officials: Håvard O Skjerven, Principal Investigator — Oslo University Hospital
Locations (9):
- Norway (9):
  - Ålesund Hospital Trust, Ålesund
  - Haukeland University Hospital, Bergen
  - Nordlandssykehuset Bodø, Bodø
  - Østfold Hospital Trust, Grålum
  - Akershus University Hospital, Lørenskog
  - Oslo University of Oslo, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of Northern Norway, Tromsø
  - St. Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No